CLINICAL TRIAL: NCT04884685
Title: A Randomized, Double-Blinded, Placebo-Controlled, Phase Ⅱb Clinical Trial, to Evaluate the Safety of the Inactivated SARS-CoV-2 Vaccine (Vero Cell) in Healthy Population Aged From 3 to 17 Years.
Brief Title: Safety of an Inactivated SARS-CoV-2 Vaccine (CoronaVac) in Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sinovac Life Sciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sinovac Biotech Co., Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PRO-nCOV-2001
Record Dates: First submitted 2021-05-07; First posted 2021-05-13 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2021-05

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — sinovac COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participant will receive two doses of medium dosage inactivated SARS-CoV-2 vaccine . Vaccine will given by intramuscular injection on day 0 and day 28.
  Interventions: Biological: SARS-CoV-2 Inactivated Vaccine
- Control Group (Placebo Comparator): Placebo will receive two doses of placebo. The placebo will given by intramuscular injection on day 0 and day 28.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 Inactivated Vaccine — 600SU inactivated virus in 0·5 mL of aluminium hydroxide solution per injection
  Other Names: CoronaVac
  Arms: Experimental Group
Biological: Placebo — aluminium hydroxide solution only
  Arms: Control Group

SUMMARY:
This study is a randomized, double-blinded, placebo-controlled, phase Ⅱb clinical trial of an inactivated SARS-CoV-2 vaccine (CoronaVac) manufactured by Sinovac Life Sciences Co. , Ltd.The purpose of this study is to evaluate the safety of the SARS-CoV-2 Inactivated vaccine in healthy children and adolescents aged 3-17 years.

DETAILED DESCRIPTION:
This study is a randomized, double-blinded, placebo-controlled,phase Ⅱb clinical trial in children and adolescents aged 3-17 years. The experimental vaccine and placebo were both manufactured by Sinovac Life Sciences Co. , Ltd. A total of 500 subjects will be enrolled, including 100 children aged 3-5 years, 200 children aged 6-11 years and 200 adolescents aged 12-17 years. Each age group will be randomly divided into two groups in a 3:1 ratio and received two doses of experimental vaccine or placebo on on day 0 and day 28.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children and adolescents aged 3-17 years;
* The subjects and/or guardians can understand and voluntarily sign the informed consent form (For subjects aged 8-17 years, both subjects and guardians need to sign the informed consent form);
* Proven legal identity.

Exclusion Criteria:

* Travel history / residence history of communities with case reports within 14 days;
* History of contact with a SARS-CoV-2 infection (positive in nucleic acid test) within 14 days;
* Have contacted patients with fever or respiratory symptoms from communities with case reports within 14 days;
* Two or more cases of fever and / or respiratory symptoms in a small contact area of volunteers, such as home, office etc. within 14 days;
* History of SARS-CoV-2 infection;
* History of asthma, history of allergy to the vaccine or vaccine components, or serious adverse reactions to the vaccine, such as urticaria, dyspnea, and angioedema;
* Congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Autoimmune disease or immunodeficiency / immunosuppression;
* Severe chronic diseases, severe cardiovascular diseases, hypertension and diabetes that cannot be controlled by drugs, liver or kidney diseases, malignant tumors, etc.;
* Severe neurological disease (epilepsy, convulsions or convulsions) or mental illness;
* Thyroid disease or history of thyroidectomy, spleenlessness, functional spleenlessness, spleenlessness or splenectomy resulting from any condition;
* Diagnosed abnormal blood coagulation function (eg, lack of blood coagulation factors, blood coagulopathy, abnormal platelets) or obvious bruising or blood coagulation;
* Immunosuppressive therapy, cytotoxic therapy, inhaled corticosteroids (excluding allergic rhinitis corticosteroid spray therapy, acute noncomplicated dermatitis superficial corticosteroid therapy) in the past 6 months;
* History of alcohol or drug abuse;
* Acute diseases or acute exacerbation of chronic diseases in the past 7 days;
* Receipt of blood products within in the past 3 months;
* Receipt of other investigational drugs in the past 30 days;
* Receipt of attenuated live vaccines in the past 14 days;
* Receipt of inactivated or subunit vaccines in the past 7 days;
* Axillary temperature >37.0°C;
* Already pregnant (including a positive urine pregnancy test) or are breastfeeding, planning to get pregnant within 3 months;
* According to the investigator's judgment, the subject has any other factors that are not suitable for participating in the clinical trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-28 after each dose
  Incidence rate of adverse reactions occured from the beginning of the vaccination to 28 days after the second dose.

SECONDARY OUTCOMES:
Safety index-incidence of adverse reactions | Day 0-7 after each dose vaccination
  Incidence rate of adverse reactions within 7 days after each dose
Safety index-incidence of serious adverse events | From the beginning of the vaccination to 6 months after the second dose vaccination
  Incidence rate of serious adverse events from the beginning of the vaccination to 6 months after the second dose vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Yuliang Zhao, Master, Principal Investigator — Hubei Provincial Center for Disease Control and Prevention
Locations (1):
- Zanhuang county Center for Disease Control and Prevention, Shijiazhuang, Hebei, China